CLINICAL TRIAL: NCT01957618
Title: The Follow-up Study of Chronic Hepatitis B Patients With Liver Cirrhosis Receiving Anti-HBV Therapy
Acronym: CTEAM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201110057RC
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis B Virus-Related Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment group: liver cirrhosis group who received indefinite anti-viral treatment
- Historical control group: Liver cirrhotic patients who were enrolled before 2004 and did not receive treatment during the follow-up

SUMMARY:
Hepatitis B virus (HBV) infection is a global health problem, especially in the endemic area like Taiwan, where there are more than 3 million chronic hepatitis B carriers. Patients with chronic HBV infection are at increased risk of developing cirrhosis, which may have disastrous complications, including hepatic decompensation, and hepatocellular carcinoma (HCC). The liver cirrhosis related complications accounts for the 8th leading cause of deaths in Taiwan; whereas, the HCC is the 2nd leading cause of deaths among all cancers. Therefore, it is prudent to develop strategies to prevent or halt the progression of liver cirrhosis.

For HBV patients who have already had cirrhosis, the main treatment objective is to reduce their risk of complications. A large-scale multicenter clinical trial showed that viral suppression using lamivudine in patients with advanced fibrosis effectively decreases the risk of HCC and liver-related complications. This study highlights the importance to treat HBV-related cirrhosis patients; however, several issues remain to be addressed.

The first issue is that this clinical trial only enrolled patients with positive HBeAg or HBV-DNA level >1.4 x105 IU/mL. However, the current recommended threshold for cirrhotic patients to start anti-viral treatment is 2000 IU/mL. Whether anti-HBV therapy benefits cirrhotic patients in this level is still unclear. Second, lamivudine was used in this clinical trial; however, the high resistant rate of lamivudine during treatment probably lowers its protective effect against HCC. Whether a more potent anti-HBV agent with extremely low resistance profile, entecavir, is more beneficial to HBV-related cirrhotic patients is also unclear.

The Bureau of National Health Institute launched the reimbursement program for anti-HBV therapy since 2003 and extended this program to cirrhotic patients with HBV DNA level > 2000 IU/mL for long-term use since Aug, 2010. Taking this advantage, we may explore the above-mentioned clinical questions more easily.

To address these issues, we will first retrospectively collect a cohort of HBV-related cirrhosis patients. All the patients will be enrolled from the time before oral anti-HBV therapy is widely used. We will determine their baseline serum HBV-DNA levels using the stored sera and enrolled those with baseline HBV-DNA levels higher than 2000 IU/mL as our historical controls. Second, we will enroll a retrospective cohort of HBV-related cirrhotic patients from 2008 who had HBV-DNA levels higher than 2000 IU/mL and received indefinite therapy of entecavir. By comparing these two cohorts, we will be able to clarify whether indefinite viral suppression by entecavir is beneficial for the cirrhotic patients.

With comprehensive analysis, we wish to document that re-setting the risk level of HBV DNA from 140,000 IU/mL to 2,000 IU/mL is more beneficial for HBV-related cirrhotic patients and long-term entecavir does lower the risk of HCC further. These lines of evidence will assist in delivering appropriate and more aggressive treatment for these high-risk patients.

ELIGIBILITY:
Inclusion Criteria for treatment group:

1. Age older than 20 years old.
2. HBsAg (+) > 6 months
3. Baseline serum HBV DNA ≧ 2000 IU/mL (10,000 copies/mL)
4. Liver cirrhosis (Child A) before or at enrollment, diagnosed by 1). Liver biopsy（Metavir F4 or Ishak > F5） or 2). Ultrasonographic evidence of cirrhosis with signs of portal hypertension (splenomegaly or presence of esophageal or gastric varices)
5. Receiving long-term anti-HBV therapy

Inclusion Criteria for control group:

1. Age older than 20 years old.
2. HBsAg (+) > 6 months
3. Baseline serum HBV DNA ≧ 2000 IU/mL (10,000 copies/mL)
4. Liver cirrhosis (Child A) before or at enrollment, diagnosed by 1). Liver biopsy（Metavir F4 or Ishak > F5） or 2). Ultrasonographic evidence of cirrhosis with signs of portal hypertension (splenomegaly or presence of esophageal or gastric varices)
5. without receiving treatment

Exclusion Criteria:

1. . Co-infection of HCV (anti-HCV (+)) or HIV
2. . Alcoholism (alcohol consumption > 20 gm/day)
3. . Serological evidence suggestive of autoimmune hepatitis, primary biliary cirrhosis, Wilson's disease and hemochromatosis
4. . Liver decompensation (Child-Pugh classification of B or C)
5. . Evidence of HCC at study entry
6. . Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
hepatocellular carcinoma | within a 10-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215